CLINICAL TRIAL: NCT00647049
Title: Freiburg ZNS-NHL Study: Therapy for Patients With Primary Non-Hodgkin Lymphoma of the CNS - Sequential High Dosage Chemotherapy With Autologous Peripheral Blood Stem Cell Plantation
Brief Title: Freiburg ZNS-NHL Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Dr. G. Illerhaus, University Hospital Freiburg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZNS-00465
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Primary Non Hodgkin Lymphoma of the Central Nervous System
MeSH Terms: interventions — Methotrexate; Rituximab; Cytarabine; Thiotepa; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): first diagnosis of PCNSL: combined chemotherapy with methotrexate
  Interventions: Drug: methotrexate; Drug: Rituximab; Drug: Cytarabine; Drug: Thiotepa; Drug: Carmustin
- B (Experimental): Patients with relapse or progressive disease of PCNSL after methotrexate containing chemotherapy
  Interventions: Drug: Rituximab; Drug: Cytarabine; Drug: Thiotepa; Drug: Carmustin

INTERVENTIONS:
Drug: methotrexate — 8000mg/m2 i.v., max. 2 cycles
  Other Names: MTX
  Arms: A
Drug: Rituximab — 375mg/m2, max. 8 times
Drug: Cytarabine — 3000mg/m2 die i.v., 2 days (max. 2 cycles)
  Other Names: Arabinoside
Drug: Thiotepa — 40mg/m2 i.v. (max. 2 cycles) 2 x 5mg/kg/die i.v. for 2 days
Drug: Carmustin — 400mg/m2 i.v. for 1 day
  Other Names: BCNU; Bis-Chlorethyl-Nitrosourea

SUMMARY:
The purpose of this study is to determine whether combined chemotherapy [rituximab plus high dosage methotrexate (max. 2 cycles) followed by arabinoside/thiotepa (max. 2 cycles) followed by high dosage carmustin/thiotepa] followed by peripheral blood stem cell transplantation is effective in the treatment of cerebral Non Hodgkin lymphoma [PCNSL].

ELIGIBILITY:
Inclusion Criteria:

* group A: first diagnosis of PCNSL, histologically confirmed
* group B: relapse or progression of PCNSL after MTX containing chemotherapy
* age 18 - 65 years
* not legally incompetent, physically or mentally incapable of giving consent
* written signed and dated informed consent of the legal representative and - if possible - of the patient

Exclusion Criteria:

* manifestations of further lymphoma outside the CNS
* sero-positive for HIV
* severe pulmonary, cardiac, hepatic, renal impairment
* neutrophil count < 2.000/µl, platelet count < 100.000/µl
* pulmonary disease with IVC < 55%, DLCO < 40%
* cardiac ejection fraction < 50%, uncontrolled malign arrhythmia
* creatinine > 1,5 mg% or creatinine-clearance < 50ml/min
* bilirubin > 2mg/dl
* ascites or pleural effusion (> 500ml)
* pregnancy o r lactation
* women with childbearing potential without sufficient contraception
* participation in another clinical trial within the last 30 days prior to the begin or parallel to this study
* known or current drug or alcohol abuse
* known hypersensitivity against methotrexate, cytarabine, thiotepa, BCNU rituximab, leukovorin, dexamethasone, neupogen and neulasta.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2007-01; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 30 days after blood stem cell transplantation

SECONDARY OUTCOMES:
Duration of response | within 5 years
Overall survival time | within 5 years
Neuropsychological state according to Mini-Mental State | within 5 years
Neuropsychological assessment (digit span, Hopkins verbal Learning Test-Revised, Trials 1-3, Brief Test of Attention, Trial Making Test, Grooved Pegboard, 6. HVLT-R , EORTC L C30 , EORTC BN20) | within 5 years
(Serious) adverse events ([S]AEs) | within 30 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Finke, Prof. Dr., Principal Investigator — University Medical Center Freiburg, Dept. of Internal Medicine I - Hematology and Oncology
Locations (1):
- University Hospital Freiburg, Freiburg im Breisgau, Germany

REFERENCES:
- [Background] Illerhaus G, Marks R, Ihorst G, Guttenberger R, Ostertag C, Derigs G, Frickhofen N, Feuerhake F, Volk B, Finke J. High-dose chemotherapy with autologous stem-cell transplantation and hyperfractionated radiotherapy as first-line treatment of primary CNS lymphoma. J Clin Oncol. 2006 Aug 20;24(24):3865-70. doi: 10.1200/JCO.2006.06.2117. Epub 2006 Jul 24. PMID 16864853
- [Derived] Kasenda B, Ihorst G, Schroers R, Korfel A, Schmidt-Wolf I, Egerer G, von Baumgarten L, Roth A, Bloehdorn J, Mohle R, Binder M, Keller U, Lamprecht M, Pfreundschuh M, Valk E, Fricker H, Schorb E, Fritsch K, Finke J, Illerhaus G. High-dose chemotherapy with autologous haematopoietic stem cell support for relapsed or refractory primary CNS lymphoma: a prospective multicentre trial by the German Cooperative PCNSL study group. Leukemia. 2017 Dec;31(12):2623-2629. doi: 10.1038/leu.2017.170. Epub 2017 May 31. PMID 28559537
- [Derived] Illerhaus G, Kasenda B, Ihorst G, Egerer G, Lamprecht M, Keller U, Wolf HH, Hirt C, Stilgenbauer S, Binder M, Hau P, Edinger M, Frickhofen N, Bentz M, Mohle R, Roth A, Pfreundschuh M, von Baumgarten L, Deckert M, Hader C, Fricker H, Valk E, Schorb E, Fritsch K, Finke J. High-dose chemotherapy with autologous haemopoietic stem cell transplantation for newly diagnosed primary CNS lymphoma: a prospective, single-arm, phase 2 trial. Lancet Haematol. 2016 Aug;3(8):e388-97. doi: 10.1016/S2352-3026(16)30050-3. Epub 2016 Jul 13. PMID 27476790